CLINICAL TRIAL: NCT03375814
Title: The Effect of Crocina on The Cellular Immune Responses in Patients With Osteoarthritis as Randomized, Double-blind and Placebo Controlled
Brief Title: Evaluation Effect of Crocina on The Cellular Immune Responses in Osteoarthritis Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shariati Jaleh, Dr. Tafaghodi Mohsen, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 931577
Record Dates: First submitted 2017-10-12; First posted 2017-12-18 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Osteoarthritis, Knee
Keywords: Crocin, osteoarthritis, Inflammation, IL-17,T-helper,T-reg
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Inflammation | interventions — crocin; Control Groups

STUDY DESIGN:
Intervention Model Description: Osteoarthritis patients who have age between 40 to 75 years old will be selected; Based on radiographic images of patients the severity of joints damage will get detailed and they will be placed in between grade 2 and grade 3 in terms of gradation; these patients will be not located underwent surgery; Patients will complete WOMAC and KOOS questionnaires to obtain some information such as following items; They will be no history of injury; they will not have diabetic disorders, rheumatism and kidney disease, osteonecrosis, gout; they will not have a long history anti-inflammatory drugs consumption; They will not have individuals with insufferable jobs carrying heavy loads; Patients will not have the Body Mass Index (BMI) of 30 or more
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The group that takes the main drug. They received the conventional treatment group and crocin.
  Interventions: Drug: Crocin
- Placebo group (Placebo Comparator): The group that takes the Placebo.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Crocin — This group (osteoarthritic patients) can receive crocin with conventional therapy
  Other Names: Test group
  Arms: Experimental group
Drug: Placebo Oral Tablet — The group that takes Placebo Oral Tablet. They received the conventional treatment and Placebo Pills..
  Other Names: Control group
  Arms: Placebo group

SUMMARY:
The effect of Crocina on the production of IL-4, IL-1 bet, IL-17, IL-10 and TGF-beta: The effect of crocina on gene expression of transcription factors T-bet, GATA-3. FOXP3, ROR-γt,; The effect of helper T cells type one and two, regulatory T cells and T helper type 17 cells; the effect of crocina on the reduction of pain and joint inflammation. Design: Randomized, Double-blind and Placebo controlled; Study population: Patients with Osteoarthritis; Volume: 40 persons; Method: Osteoarthritis patients will be divided into two groups according to age and sex; Crocina tablets will be prescribed to the first group a tablet 15 mg daily along with conventional Medicines; Placebo tablets will be prescribed to the second group along with the conventional medicines; Blood sampling of patients will be done before drug administering and four months after treatment. Major Inclusion Criteria: Osteoarthritis patients with age 40-75 years; The severity of joint damage between grade 2 and 3; Patients without history of injury; Patients with body mass index less than 30. Major Exclusion Criteria: Osteoarthritis patients with age 40-75 years; The severity of joint damage in grade one and four; Patients with history of injury and body mass index 30 or more. Intervention: Treatment with prescription of drug at dose of 15 mg daily crocin in the study group and placebo in the control group. Time: 4 months; Main outcome Measures: Osteoarthritis, Pain, Inflammation, Crocina, IL-4, IL-1 beta, IL-17, IL-10, TGF- beta, Cell surface protein CD127, The expression of T-bet, GATA-3, FOXP3, ROR-γt and the number of Th1, Th2, T-regulatory and Th17.

DETAILED DESCRIPTION:
The effect of crocina on the production of IL-4, IL-1β, IL-17, IL-10 and TGF-β by ELISA assay;The effect of crocina on gene expression of transcription factors T-bet, GATA3, FOXP3, ROR-γt by Real-Time PCR; The effect of crocina on number of helper T cells type one and two, regulatory T cells and T helper type 17 cells by Flow Cytometry analysis; The effect of crocina on the reduction of pain and joint inflammation by WOMAC osteoarthritis index, vas score pain and CRP, ESR diagnostic tests . Design: Randomized, Double-blind and Placebo controlled; Study population: Patients with Osteoarthritis; Volume: 40 persons; Method: Osteoarthritis patients will be divided into two groups according to age and sex; Crocina tablets will be prescribed to the first group a tablet 15 mg daily along with the conventional medicines. 30 pills of crocina or placebo in cans quite similar and be encoded with Excel Software will be given to the patients completely random; The distributor and the patient will have no knowledge of the contents of the cans; After the end of each month, the patients will receive similar to their previous code. Blood sampling of patients will be done before drug administering and four months after the treatment. Major Inclusion Criteria: Osteoarthritis patients with age 40 to 75 years; The severity of joint damage between grade 2 and 3; Patients without history of injury; Patients with the Body Mass Index (BMI) less than 30. Major Exclusion Criteria: Osteoarthritis patients with age less than 40 and more than 75; The severity of joint damage in the grade one and four; Patients with history of injury and body mass index 30 or more. Intervention: Treatment with prescription of drug at dose of 15 mg daily crocin in the study group and placebo in the control group; Time: 4 months. Main Outcome Measures: Osteoarthritis, Pain, Inflammation, Crocin, IL-4, IL-1 beta, IL-17, IL-10, TGF-beta, Cell surface CD127, The expression of T-bet; GATA3; FOXP3; RORgt and the number of Th1, Th2, T-regulatory and Th17

ELIGIBILITY:
Inclusion Criteria:

Osteoarthritis patients must have

* Aged 40 to 75.
* The severity of joint damage between grade 2 and grade 3 based on radiographic images.
* No history of joint surgery.
* No history of injury.
* No diabetic disorders.
* No rheumatism.
* No kidney disease.
* No osteonecrosis and gout.
* No long history of anti-inflammatory drugs consumption.
* No insufferable jobs;
* The Body Mass Index (BMI) of 30 or less.

Exclusion Criteria:

Osteoarthritis patients should not have:

* Aged less than 40 and more than 75
* With the severity of joint damage of the in grade 1 and grade 4 based on radiographic images.
* With history of joint surgery.
* With history of injury
* With diabetic disorders, rheumatism, kidney disease, osteonecrosis and gout.
* With long history of anti-inflammatory drugs consumption.
* Having insufferable jobs.
* With a BMI of 30 or more.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-07-20 (Actual); Primary Completion 2018-03-02 (Estimated); Study Completion 2018-07-30 (Estimated)

PRIMARY OUTCOMES:
Radiographic report from knee | 15 minute
  Patients suffering from osteoarthritis are classified in grades 1 to 4 and grades 2 and 3 will be enter to study.

CONTACTS AND LOCATIONS:
Locations (1):
- Jaleh Shariati sarabi, Mashhad, Razavi Khorasan Province, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mohebbi M, Atabaki M, Tavakkol-Afshari J, Shariati-Sarabi Z, Poursamimi J, Mohajeri SA, Mohammadi M. Significant Effect of Crocin on the Gene Expression of MicroRNA-21 and MicroRNA-155 in Patients with Osteoarthritis. Iran J Allergy Asthma Immunol. 2022 Jun 18;21(3):322-331. doi: 10.18502/ijaai.v21i3.9805. PMID 35822682